CLINICAL TRIAL: NCT06009900
Title: Safety and Efficacy of Low-intensity Laser Therapy in the Treatment of Chronic Musculoskeletal Pain: a Multicenter Randomized Controlled Trail
Brief Title: Safety and Efficacy of Low-intensity Laser Therapy in the Treatment of Chronic Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Shanxi Bethune Hospital (Other); Second Hospital of Shanxi Medical University (Other); Shanxi Provincial People's Hospital (Other Government); China Resources WISCO General Hospital (Unknown); LinFen People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJ-IRB20230796
Record Dates: First submitted 2023-08-07; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Pain, Chronic
Keywords: Chronic musculoskeletal pain; Low intensity laser therapy; Non-steroidal drugs
MeSH Terms: conditions — Chronic Pain | interventions — Celecoxib; Population Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-steroidal drug (Celecoxib) group (Active Comparator): Oral Celecoxib 200mg/time, twice a day, for three consecutive weeks.
  Interventions: Drug: Non-steroidal drug (Celecoxib) group
- Weak laser treatment group (Experimental): Low intensity laser treatment: Both patients and doctors wear goggles during the irradiation process. Using 810nm (infrared)/658nm (red) dual wavelength output for direct skin contact point irradiation, the maximum output power is 100mW (red)/60mW (infrared). Select the treatment site based on the patient's anatomical positioning (muscle and tendon attachment points, nerve distribution aggregation points) and/or pain points, and perform spot laser irradiation. Low intensity laser treatment process: Treat once a day for 15 minutes each time, with 5 consecutive days of treatment and 2 days of rest per week. The patient received a total of 3 weeks (15 times) of low intensity laser treatment.
  Interventions: Device: Low intensity laser treatment

INTERVENTIONS:
Device: Low intensity laser treatment — Low intensity laser treatment: Both patients and doctors wear goggles during the irradiation process. Using 810nm (infrared)/658nm (red) dual wavelength output for direct skin contact point irradiation, the maximum output power is 100mW (red)/60mW (infrared). Select the treatment site based on the patient's anatomical positioning (muscle and tendon attachment points, nerve distribution aggregation points) and/or pain points, and perform spot laser irradiation. Low intensity laser treatment process: Treat once a day for 15 minutes each time, with 5 consecutive days of treatment and 2 days of rest per week. The patient received a total of 3 weeks (15 times) of low intensity laser treatment.
  Arms: Weak laser treatment group
Drug: Non-steroidal drug (Celecoxib) group — Oral Celecoxib 200mg/time, twice a day, for three consecutive weeks.
  Arms: Non-steroidal drug (Celecoxib) group

SUMMARY:
This study is a multicenter, prospective, randomized, controlled research design. This study takes classic NSAIDs treatment as a control, and it will take patients' pain relief, functional improvement, sleep quality improvement, and adverse reactions as the main and secondary evaluation indicators to explore the safety and effectiveness of weak laser treatment of chronic musculoskeletal pain, determining the dominant disease in the treatment of Chronic pain.

DETAILED DESCRIPTION:
Research purpose:

Chronic musculoskeletal pain is the most common clinical Chronic pain. Non-steroidal drugs are the most commonly used therapeutic drugs, but their effects on improving the body function are limited. At present, the pain diagnosis and treatment guidelines recommend that non-drug treatment should be used as a first-line treatment measure. Low intensity laser therapy can alleviate chronic musculoskeletal pain through multiple effects such as anti-inflammatory, promoting blood circulation, and promoting tissue repair. However, a large number of high-quality clinical studies are still needed to confirm its effectiveness. In view of this, this study aims to investigate the safety and effectiveness of dual wavelength weak laser therapy for chronic musculoskeletal pain independently developed in China, in order to clarify the clinical application value of this technology.

Research protocol:

This study is an intervention study. The participants will be assigned to different treatment groups (drug therapy group or low intensity laser therapy) to receive corresponding treatment. At the end of treatment and 1, 2, and 3 months after treatment, the researchers will evaluate treatment efficacy through a questionnaire survey.

This study will (1) compare the degree of pain relief, functional improvement, sleep quality, quality of daily life, and incidence of adverse reactions in patients with chronic musculoskeletal pain after receiving weak laser therapy and NSAIDs treatment; (2) study the analgesic effect of low intensity laser therapy on different types of chronic musculoskeletal pain, and determine the advantageous disease types for this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Chronic musculoskeletal pain (including cervical spondylosis, periarthritis of shoulder, osteoarthritis, back muscle Fasciitis, lumbar disc herniation) was diagnosed, and the pain lasted for more than 3 months;
3. The degree of pain before treatment was mild to moderate (NRS score<7 points);
4. Can cooperate in completing consultation and scale evaluation;
5. Sign an informed consent form.

Exclusion Criteria:

1. Previous spinal surgery or severe spinal diseases (such as fractures, tumors, inflammation, and infectious diseases);
2. Suffering from serious systemic diseases, including liver and kidney dysfunction, cardio cerebral, vascular disease, decompensated metabolic syndrome;
3. Serious skin diseases (skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis, lupus, Hives);
4. Suffering from mental disorders, intellectual disabilities, epilepsy and other diseases;
5. Moderate to severe depressive state;
6. Have a history of drug abuse, drug abuse, and alcohol abuse;
7. Individuals with contraindications to NSAIDs or laser therapy;
8. Pregnant women;
9. Recently participated in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness | the end of treatment (day21)
  At the end of treatment (day21), the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 30% in total patients. This proportion is defined as the treatment effectiveness rate.

SECONDARY OUTCOMES:
the proportion of patients with a decrease in NRS score of ≥ 30% 1 month after treatment | 1 month after treatment
  1 month after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 30% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 30% 2 months after treatment | 2 months after treatment
  2 months after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 30% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 30% 3 months after treatment | 3 months after treatment
  3 months after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 30% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 50% at the end of treatment | the end of treatment (day21)
  At the end of treatment (day21), the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 50% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 50% 1 month after treatment | 1 month after treatment
  1 month after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 50% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 50% 2 months after treatment | 2 months after treatment
  2 months after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 50% in total patients. This proportion is defined as the treatment effectiveness rate.
the proportion of patients with a decrease in NRS score of ≥ 50% 3 months after treatment | 3 months after treatment
  3 months after treatment, the pain NRS (0, no pain; 10, worst pain imaginable) of patients are collected. These data are used to calculate the percentage of the difference between them and pain NRS of patients before treatment, relative to the latter. Then, this study calculates the proportion of patients with a decrease in NRS score of ≥ 50% in total patients. This proportion is defined as the treatment effectiveness rate.
NRS at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, Numerical Rating Scale (NRS) (0, no pain; 10, worst pain imaginable) of pain is collected.
NRS 1 month after treatment | 1 month after treatment
  1 month after treatment, Numerical Rating Scale (NRS) (0, no pain; 10, worst pain imaginable) of pain is collected.
NRS 2 months after treatment | 2 months after treatment
  2 months after treatment, Numerical Rating Scale (NRS) (0, no pain; 10, worst pain imaginable) of pain is collected.
NRS 3 months after treatment | 3 months after treatment
  3 months after treatment, Numerical Rating Scale (NRS) (0, no pain; 10, worst pain imaginable) of pain is collected.
BPI at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, Brief Pain Inventory (BPI) (11-Point scale, 0 = does not interfere, 10 = completely interferes; Higher score = greater pain or interference of pain with activities, sleep, and negative mood.) is collected.
BPI 1 month after treatment | 1 month after treatment
  1 month after treatment, Brief Pain Inventory (BPI) (11-Point scale, 0 = does not interfere, 10 = completely interferes; Higher score = greater pain or interference of pain with activities, sleep, and negative mood.) is collected.
BPI 2 months after treatment | 2 months after treatment
  2 months after treatment, Brief Pain Inventory (BPI) (11-Point scale, 0 = does not interfere, 10 = completely interferes; Higher score = greater pain or interference of pain with activities, sleep, and negative mood.) is collected.
BPI 3 months after treatment | 3 months after treatment
  3 months after treatment, Brief Pain Inventory (BPI) (11-Point scale, 0 = does not interfere, 10 = completely interferes; Higher score = greater pain or interference of pain with activities, sleep, and negative mood.) is collected.
RMDQ at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, Roland Morris Disability Questionnaire (RMDQ) (Scores 0 to 24, higher score, indicates greater activity limitation) is collected.
RMDQ 1 month after treatment | 1 month after treatment
  1 month after treatment, Roland Morris Disability Questionnaire (RMDQ) (Scores 0 to 24, higher score, indicates greater activity limitation) is collected.
RMDQ 2 months after treatment | 2 months after treatment
  2 months after treatment, Roland Morris Disability Questionnaire (RMDQ) (Scores 0 to 24, higher score, indicates greater activity limitation) is collected.
RMDQ 3 months after treatment | 3 months after treatment
  3 months after treatment, Roland Morris Disability Questionnaire (RMDQ) (Scores 0 to 24, higher score, indicates greater activity limitation) is collected.
PSQI 3 months after treatment | 3 months after treatment
  3 months after treatment, Pittsburgh Sleep Quality Index (PSQI) (Higher score = better sleep quality) is collected.
PSQI 2 months after treatment | 2 months after treatment
  2 months after treatment, Pittsburgh Sleep Quality Index (PSQI) (Higher score = better sleep quality) is collected.
PSQI 1 month after treatment | 1 month after treatment
  1 month after treatment, Pittsburgh Sleep Quality Index (PSQI) (Higher score = better sleep quality) is collected.
PSQI at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, Pittsburgh Sleep Quality Index (PSQI) (Higher score = better sleep quality) is collected.
EQ-5D at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, EuroQoL-5D (EQ-5D) (Each item, 3 levels 1 = no problem, 2 = some problem, 3 = extreme problem. Range, 0 = worst imaginable, 100 best imaginable health state) is collected.
EQ-5D 1 month after treatment | 1 month after treatment
  1 month after treatment, EuroQoL-5D (EQ-5D) (Each item, 3 levels 1 = no problem, 2 = some problem, 3 = extreme problem. Range, 0 = worst imaginable, 100 best imaginable health state) is collected.
EQ-5D 2 months after treatment | 2 months after treatment
  2 months after treatment, EuroQoL-5D (EQ-5D) (Each item, 3 levels 1 = no problem, 2 = some problem, 3 = extreme problem. Range, 0 = worst imaginable, 100 best imaginable health state) is collected.
EQ-5D 3 months after treatment | 3 months after treatment
  3 months after treatment, EuroQoL-5D (EQ-5D) (Each item, 3 levels 1 = no problem, 2 = some problem, 3 = extreme problem. Range, 0 = worst imaginable, 100 best imaginable health state) is collected.
HADS 3 months after treatment | 3 months after treatment
  3 months after treatment, Hospital Anxiety and Depression Scale (HADS) (Total score can be used as a measure of global negative affect. Score 8 to 10 = mild, 11 to 15 = moderate, ≥ 16 = severe) is collected.
HADS 2 months after treatment | 2 months after treatment
  2 months after treatment, Hospital Anxiety and Depression Scale (HADS) (Total score can be used as a measure of global negative affect. Score 8 to 10 = mild, 11 to 15 = moderate, ≥ 16 = severe) is collected.
HADS 1 month after treatment | 1 month after treatment
  1 month after treatment, Hospital Anxiety and Depression Scale (HADS) (Total score can be used as a measure of global negative affect. Score 8 to 10 = mild, 11 to 15 = moderate, ≥ 16 = severe) is collected.
HADS at the end of treatment (day21) | the end of treatment (day21)
  At the end of treatment, Hospital Anxiety and Depression Scale (HADS) (Total score can be used as a measure of global negative affect. Score 8 to 10 = mild, 11 to 15 = moderate, ≥ 16 = severe) is collected.

OTHER OUTCOMES:
Adverse reactions | during treatment (From start of treatment until the end of treatment or date when patient cannot continue the current treatment, whichever came first, assessed up to 21 days)
  Adverse reactions, such as non-steroidal drugs-associated adverse reaction, weak laser-related skin damage
Adverse reactions | the end of treatment (day21)
  Adverse reactions, such as non-steroidal drugs-associated adverse reaction, weak laser-related skin damage
Adverse reactions | 1 month after treatment
  Adverse reactions, such as non-steroidal drugs-associated adverse reaction, weak laser-related skin damage
Adverse reactions | 2 months after treatment
  Adverse reactions, such as non-steroidal drugs-associated adverse reaction, weak laser-related skin damage
Adverse reactions | 3 months after treatment
  Adverse reactions, such as non-steroidal drugs-associated adverse reaction, weak laser-related skin damage
NRS before treatment | before treatment
  Before treatment, pain NRS (0, no pain; 10, worst pain imaginable) is collected.
BPI before treatment | before treatment
  Before treatment, BPI (11-Point scale, 0 = does not interfere, 10 = completely interferes; Higher score = greater pain or interference of pain with activities, sleep, and negative mood.) is collected.
RMDQ before treatment | before treatment
  Before treatment, RMDQ (Scores 0 to 24, higher score, indicates greater activity limitation) is collected.
PSQI before treatment | before treatment
  Before treatment, PSQI (Higher score = better sleep quality) is collected.
EQ-5D before treatment | before treatment
  Before treatment, EQ-5D (Each item, 3 levels 1 = no problem, 2 = some problem, 3 = extreme problem. Range, 0 = worst imaginable, 100 best imaginable health state) is collected.
HADS before treatment | before treatment
  Before treatment, HADS (Total score can be used as a measure of global negative affect. Score 8 to 10 = mild, 11 to 15 = moderate, ≥ 16 = severe) is collected.
Patient basic information | before treatment
  Patient basic information includes gender, age, marital status, education level (high school and below, university, graduate), occupational status (employment/education/retirement), height, weight, BMI, smoking history, and past history; Clinical characteristics related to the disease include history of low back pain (time of Chronic pain (years), number of acute attacks, time of this attack), and history of treatment of low back pain

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - China Resources & WISCO General Hospital, Wuhan, Hubei
  - LinFen People's Hospital, Linfen, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi